CLINICAL TRIAL: NCT01476579
Title: Diagnostic Accuracy of New Generation Low-dose CT Coronary Angiography
Brief Title: Comparison of Low-radiation Dose CT Angiography With Invasive Coronary Angiography in Stable Coronary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/123
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary CT; Sensitivity; Specificity; Radiation; Tomography, X-Ray Computed; Coronary angiography
MeSH Terms: conditions — Coronary Artery Disease; Hypersensitivity | interventions — Cardiac-Gated Single-Photon Emission Computer-Assisted Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-invasive CT coronary angiography (Other): This study is evaluating diagnostic accuracy of non-invasive CT coronary angiography with invasive coronary angiography.
  Interventions: Device: Cardiac Computer Tomography

INTERVENTIONS:
Device: Cardiac Computer Tomography — Compare Cardiac CT with reference standard wich is conventional invasive coronary angiography.

SUMMARY:
This study is evaluating the performance of modern CT coronar angiography with low radiation technique compared to conventional invasive coronar angiography. The patients recruited will already be accepted for invasive coronary angiography based on clinical presentation, ECG and biochemical parameters. An "all-comers" design to avoid selection bias and no additional B-blockers will be used prior to CT angiography. The hypothesis is that it is possible to rule out significant coronary artery disease with sensitivity > 95 % and negative predictive value > 95 % with very low radiation doses.

DETAILED DESCRIPTION:
Conventional invasive coronary angiography (CICA) is associated with few but serious complications. It is time consuming for the patient and incur costs to the health institution due to the post-procedure observation needed. Coronary computer tomography angiography (CCTA) is a good alternative to CICA to rule out coronary artery disease (CAD). Moderate to excellent sensitivity and negative predictive values have been reported with 64-slice CT angiography. The main ethical problem has been the radiation doses given to the patient during CT angiography which was high >10 millisievert(mSv). With 265 or higher slice CT machines and radiation dose reduction techniques, it is possible to evaluate coronary anatomy with radiation doses below 1 mSv. Heart rate reduction with B-blockers is in most cases not necessary with new generation CT machines but is recommended in guidelines.

800 patients already accepted for CICA based on clinical information will be scheduled to undergo CCTA prior to invasive coronary angiography. Coronary anatomy will be described according to American Heart Association (AHA) classification with 17 segment analysis. The main purpose of the study is to achieve high sensitivity and high negative predictive value with CT angiography. Radiation doses in relation to gender and body mass index (BMI) will be monitored. In addition we will measure coronary calcification (Agatson score) and look at any association to the Vitamin D and calcium metabolism. Patient reported quality of life evaluation with validated questionnaires and long term follow up (5 and 10 years) regarding clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. 800 Patients who are scheduled to undergo conventional invasive coronary angiogram will be recruited at the University hospital of North Norway, Tromsø.

Exclusion Criteria:

1. Acute coronary syndrome with positive high sensitive troponin.
2. Renal failure with glomerular filtration rate (GFR) < 30
3. Contraindication to contrast medium
4. Symptomatic Tachycardia >110 or bradycardia < 40
5. Pregnancy
6. Lack of informed consent

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | 24 hours
  The results from the CT coronary angiography will be compared with the results from the conventional invasive coronary angiography which in this respect is considered the "gold standard". The sensitivity and specificity for the CT angiography regarding detection of significant coronary stenosis (ie more than 50 % lumen narrowing with the angiographic result as reference) and for revascularisation will be calculated separately.

SECONDARY OUTCOMES:
Change in quality of life and symptom score | 6 months, 1 and 3 years
  Change from baseline in quality of life and symptoms as measured with SF-12, HADS og SEATTLE will be assessed both for patients with and without significant coronary pathology with postal questionnaires at 6 months, 1 and 3 years after the CT angiography
Coronary calcium score impact on pretest coronary risk scoring and prognosis | 24 hours, 5 and 10 years
  The change in pretest probability for detection of significant stenosis and revascularisation by calcium score will be calculated in addition to prediction of 5 and 10 year fatal and non fatal cardiovascular events.
Vitamin D and other novel cardiovascular risk factors | 24 hours, 5 and 10 years
  The association of vitamin D levels (25OHD) and Single Nucleotide Polymorphism (SNP) related to vitamin D and calcium metabolism to presence of coronary plaques and their calcium content will be analysed as well as risk of fatal and non fatal coronary events. When events are registered other new novel risk markers detected in the Tromso Study will be measured in a nested case control design.
Real life radiation risk with new CT scanners and conventional invasive angiography | 24 hours
  The radiation doses will be measured independent of supplier software for both procedures and compared. Impact of risk factors on radiation dosage and image quality will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: AMJID IQBAL, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway